CLINICAL TRIAL: NCT05401227
Title: Glutamatergic Mechanisms of Psychosis and Target Engagement: Aim2
Brief Title: Glutamatergic Mechanisms: Aim2
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8299
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of three ketamine arms. with in each ketamine arm, subjects will be randomized to TS-134 or placebo for 6 total arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- High Ketamine, TS-134 (Experimental): Two administrations of ketamine 0.23 mg/kg pre post 4 days of TS-134 20 mg
  Interventions: Drug: Ketamine; Drug: Ts-134
- High ketamine, placebo (Placebo Comparator): Two administrations of ketamine 0.23 mg/kg pre post 4 days of placebo
  Interventions: Drug: Ketamine; Drug: Placebo
- Medium Ketamine, TS-134 (Experimental): Two administrations of ketamine 0.125 mg/kg pre post 4 days of TS-134 20 mg
  Interventions: Drug: Ketamine; Drug: Ts-134
- Medium Ketamine, placebo (Placebo Comparator): Two administrations of ketamine 0.125 mg/kg pre post 4 days of placebo
  Interventions: Drug: Ketamine; Drug: Placebo
- Low Ketamine, TS-134 (Experimental): Two administrations of ketamine 0.06 mg/kg pre post 4 days of TS-134 20 mg
  Interventions: Drug: Ketamine; Drug: Ts-134
- Low Ketamine, placebo (Placebo Comparator): Two administrations of ketamine 0.06 mg/kg pre post 4 days of placebo
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine during an MRI
Drug: Ts-134 — 4 days of TS-134 20 mg
  Arms: High Ketamine, TS-134; Low Ketamine, TS-134; Medium Ketamine, TS-134
Drug: Placebo — 4 days of placebo TS-134
  Arms: High ketamine, placebo; Low Ketamine, placebo; Medium Ketamine, placebo

SUMMARY:
This is a randomized, double-blind, and placebo controlled. 120 HV will be randomized to one of three ketamine arms, delivered in a bolus dose over one minute: low (0.086 mg/kg), medium (0.125 mg/kg), and high (0.23 mg/kg).

Within each ketamine arm, subjects will be randomized to 4 days of TS-134 20 mg or placebo in a 5:3 ratio (25 TS-134:15 placebo). Following an outpatient Screening Period (up to 31 days), eligible subjects will undergo an up to 5-day inpatient Treatment Period. During the study, each subject will undergo a total of two ketamine sessions: a first session during the Screening Period and a second session on Day 4 of the Treatment Period, conducted at least 7 days apart. All randomized subjects will be dosed with TS-134 or placebo daily in a fed state for 4 days during the study, titrated to 20 mg over the first 2 days.

DETAILED DESCRIPTION:
Schizophrenia (Sz) is associated with psychotic symptoms, such as hearing voices and paranoid beliefs that remain partially or fully refractory to standard antipsychotic medications for ~2/3 of patients. Alternative, glutamatergic approaches for treatment development have been proposed but have not yet led to FDA-approved medications. Moreover, several glutamate-targeted medications, such as pomaglumetad (POMA), have failed in pivotal clinical trials despite robust effectiveness in preclinical models. A major barrier to effective glutamatergic treatment development is the absence of validated measures for target engagement that can identify effective compounds and guide dose selection. Target" refers to a factor that an intervention is intended to modify, leading to improvement in symptoms, and target engagement biomarkers are a measure of the ability of the intervention to "engage" the target.

As part of the recently completed NIMH multicenter FAST-PS initiative and a parallel industry sponsored project, we evaluated ketamine-induced pharmacoBOLD (phBOLD) in healthy volunteers (HV) as a potential target engagement biomarker for development of metabotropic glutamate (mGluR2/3) agonists, as a prelude to planned studies in Sz. BOLD imaging indirectly measures brain energy, as a proxy for glutamate target engagement.

The structure of the R01 grant funding this protocol was split into three studies, specific aim (SA) 1, 2 and 3. In FAST-PS, a high dose of ketamine (0.23 mg/kg) was used in order to produce robust pharmacological effects.

Under SA1, which was conducted under IRB 8063, this dose was titrated downward in across two phBOLD sessions in HV in order to determine the lowest dose of ketamine that still produces a phBOLD response of Cohen's d≥1.5, hypothesizing that this dose would provide the best signal to noise for use in SA2. The study was conducted in groups of 10 subject per dose cohort, and the analysis supports using a low dose of 0.086 mg/kg for SA2.

SA2 experiments are modeled after our preliminary TS-134 studies. SA2 will be randomized, double-blind, and placebo controlled. 120 HV will be randomized to one of three ketamine arms: low, medium, and high. Based on SA1, the low dose will be 0.086 mg/kg. The medium dose, 0.125 mg/kg, is based the previously published mGluR2/3 target engagement study and the high dose is equal to 0.23 mg/kg, the same as in the FAST-PS study.

Within each ketamine arm, subjects will be randomized to 4 days of TS-134 20 mg or placebo in a 5:3 ratio (25 TS-134:15 placebo). Following an outpatient Screening Period (up to 31 days), eligible subjects will undergo an up to 5-day inpatient Treatment Period. During the study, each subject will undergo a total of two ketamine sessions: a first session during the Screening Period and a second session on Day 4 of the Treatment Period, conducted at least 7 days apart. All randomized subjects will be dosed with TS-134 or placebo daily in a fed state for 4 days during the study, titrated to 20 mg over the first 2 days. As before, subjects' general health and safety status will be confirmed by a phone call following discharge from the Treatment Period. Primary outcomes will be (1) suppression of the phBOLD response and (2) psychiatric symptoms after 4 days of TS-134, relative to ketamine screening session effects.

In parallel, we will evaluate sLASER MRS to interrogate the glutamate system . These additional measures will be collected at baseline, pre ketamine.

For up to the 1st 20 subjects, we will not randomize to low dose, and subjects will only receive either high or medium dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-55
2. Medically healthy, as assessed by study physician
3. Capable of understanding the study procedures and able to provide informed consent
4. Eligible men and women must agree to use a reliable method of birth control (for example, use of oral contraceptives or Norplant; a reliable barrier method of birth control diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) during the study. Women who are post-menopausal or otherwise not of childbearing potential are also eligible.

Exclusion Criteria:

1. Current or past Axis I psychiatric history (including Substance Use Disorder/Alcohol Use Disorder, with the exception of nicotine use disorder)
2. Positive urine toxicology
3. History of recreational ketamine use, recreational PCP use, or an adverse reaction to ketamine. Subjects who have participated in prior research ketamine studies will be eligible. Subjects can have infusions not more frequently than biweekly, and not more than 1/month on average, therefore subjects entering the study will need to wait one month if they had a single infusion and 6 weeks if they have had two closely spaced infusions.
4. History of first-degree relative with schizophrenia
5. Pregnancy or breast-feeding. This exclusion criterion applies only to females of child-bearing potential (not surgically sterilized and between menarche and 1 year postmenopausal). Must test negative for pregnancy at the time of screening based on a serum pregnancy test.
6. History of violence, including any history of using a gun, knife, or other weapon with intent to harm someone, as well as a more than one physical fight without a weapon after the age of 18 years old (not including fights that happen during sports competition).
7. Presence or positive history of significant medical illness, including renal problems (GFR<60), high blood pressure (defined as systolic blood pressure (SBP) > 140 or diastolic blood pressure (DBP) > 90), low blood pressure (SBP < 100, DBP < 60), orthostatic blood pressure at baseline (change in mean arterial pressure [1/3 systolic + 2/3 diastolic] of > 20%), cardiac illness, or clinically significant abnormal screening labs, as determined by the site physician.
8. Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator.
9. Presence or positive history of neurological illness, including seizures, mental retardation or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS), or history of significant head injury.
10. Metal implants, pacemaker, other metal (e.g., shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with the MR scan.
11. Medicinal patch, unless removed prior to the MR scan
12. Claustrophobia
13. Currently taking any psychotropic medication, including antidepressant medications, benzodiazepines, antipsychotic medications, mood stabilizers, anti-epileptic medications, and stimulants. We will exclude any subject who requires treatment with any psychotropic medication from one of these classes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Final PharmacoBOLD signals in pre-specified ROIs | Baseline and Day 4
  Changes in ketamine-induced PharmacoBOLD fMRI signals in pre-specified ROIs (anterior cingulate cortex) following administrations of TS-134
Brief Psychiatric Rating Scale (BPRS) | Baseline and Day 4
  Changes in BPRS scores following administrations of TS-134

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kantrowitz, MD, Principal Investigator — NYSPI
Locations (1):
- NYSPI, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH Data archive
Supporting Information: Study Protocol, ICF
Time Frame: Per NIMH Data archive regulations
Access Criteria: Qualified investigator